CLINICAL TRIAL: NCT03415399
Title: Phase 1, Open-label, Single-arm, Dose-escalation Clinical Study Evaluating the Safety and Efficacy of ET190L1 ARTEMIS™ (Anti-CD19-ARTEMIS™) in Relapsed, Refractory B Cell Lymphoma
Brief Title: Clinical Study of ET190L1 ARTEMIS™ in Relapsed, Refractory B Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eureka Therapeutics Inc. (Industry)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ETCH17CD19AR103
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Lymphoma, B-Cell
Keywords: relapsed/refractory CD19+ Lymphomas, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- i.v. arm (Experimental): ET190L1 ARTEMIS™ T cells administered by intravenous (IV) infusion
  Interventions: Biological: ET190L1 ARTEMIS™ T cells

INTERVENTIONS:
Biological: ET190L1 ARTEMIS™ T cells — Autologous T cells transduced with lentivirus encoding an anti-CD19 (ET190L1) ARTEMIS™ expression construct

SUMMARY:
This study is to determine the safety, including potential dose limiting toxicities, of ET190L1 ARTEMIS™ T cells and the duration of in vivo survival of ET190L1 ARTEMIS™ T cells in patients with relasped/refractory B-cell lymphoma. For patients with detectable disease, the study will also measure anti-tumor responses after ET190L1 ARTEMIS™ cell infusions.

DETAILED DESCRIPTION:
ET190L ARTEMIS™ is a novel chimeric T-cell therapy platform that in preclinical studies, functionally matches the efficacy of CAR T cells, but dramatically reduces the release of cytokines upon killing of target-positive tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed/refractory CD19+ B-cell lymphoma, with no effective therapy available per NCCN guidelines
* No HCV, HIV infection, no active HBV
* Liver and kidney function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) does not exceed five times the upper limit of normal range. ALT <200U / L, bilirubin <2.0 mg/ dL
* Renal function: creatinine <2.5mg / dL; Pre-treatment absolute creatinine clearance ≥50 mL / minute
* CBC: Hemoglobin ≥ 80g / L, Absolute Neutrophil Counts ≥1 × 10^9 / L, Platelets ≥50 × 10^9 / L
* Echocardiography or multiple gated angiogram (MUGA) ejection fraction> 45%
* ECOG performance status ≤2, expected survival time > 3 months per PIs opinion
* Women of childbearing age should have a negative pregnancy test and agree to use effective contraception during treatment and 1 year after the last dose.
* Had a recurrence after at least a first-line systemic treatment
* Peripheral venous access is available and no issues with apheresis for lymphocyte isolation
* Voluntarily signed informed consent form

Exclusion Criteria:

* Women in pregnancy and lactation
* Unable to perform leukapheresis and iv infusion
* With active infection
* Major organ failure
* Continuously used glucocorticoids or other immunosuppressive agents within 4 weeks
* T cell deficiency or T cells are difficult to be transduced

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 28 days up to 24 months
  Determine the safety, including potential dose limiting toxicities, of the ET190L1 ARTEMIS™ T cells. A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the ET190L1 ARTEMIS™ T-cells, which is irreversible or life threatening or CTCAE Grade 3-5. Assessed at all visits.
Toxicity profile of ET190L1 ARTEMIS™ T-cell treatment | 28 days up to 24 months
  Frequency of treatment-related adverse events that occurred at any time from the first day of infusion that are "possibly", "likely", or "definitely" related to the study, including infusion related toxicity and ET190L1 ARTEMIS™-cell T cells related toxicity. Include but not limited to: Fever, chills, nausea, vomiting, jaundice and other gastrointestinal symptoms; Fatigue, hypotension, respiratory distress; Tumor lysis syndrome; Cytokine release syndrome; Neutropenia, thrombocytopenia; Liver and kidney dysfunction. Assessed at all visits.
Tmax of serum cytokine levels | 24 weeks
  Increases or decreases in the amount of cytokine produced compared to baseline at time points measured up to 24 weeks since dosing. Cytokines as measured by Bio-Plex Multiplex Immuoassays will be presented as time to peak level.
Time to baseline for serum cytokine levels | 24 weeks
  Increases or decreases in the amount of cytokine produced compared to baseline at time points measured up to 24 weeks since dosing. Cytokines as measured by Bio-Plex Multiplex Immuoassays will be presented as Time to baseline.
AUC of serum cytokine levels | 24 weeks
  Increases or decreases in the amount of cytokine produced compared to baseline at time points measured up to 24 weeks since dosing. Cytokines as measured by Bio-Plex Multiplex Immuoassays will be presented as area under curve (AUC).
Duration of in vivo engraftment of ET190L1 ARTEMIS™ T cells | 24 months
  Number and % of ET190L1 ARTEMIS™ T cells in peripheral blood will be presented as Time to peak, Time to baseline level and the overall exposure will be presented as area under curve (AUC).

SECONDARY OUTCOMES:
Rate of disease response | 28 days to 24 months
  Rate of disease response assessed by Lugano (Chason) classification. Response rates will be estimated as the percent of patients with complete remission (CR), partial response (PR), stable disease (SD), progression disease (PD), overall survival (OS).
Anti-tumor responses | 4 months, 1 year, 2 years
  Progression free survival (PFS) and Median survival (MS) at 4 months, 1 year, 2 years
B cell depletion | 2 years
  Number and % of B cells in peripheral blood will be presented as Time to baseline level and time to recover for up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, MD, Principal Investigator — Peking University
Locations (1):
- Peking University Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No